CLINICAL TRIAL: NCT03965975
Title: (In Spanish, Spain) "Validación Clínica Mediante Estudio analítico Con Muestras de Orina Para Comparar la Eficacia y Seguridad de un Smart Device"
Brief Title: Clinical Validation Through Analytical Study With Urine Samples to Compare the Effectiveness and Security of an Intelligent Device
Acronym: STSD-2019-001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: S-There Technologies SL (Industry)
Collaborators: Biobizkaia Health Research Institute (Other Government); Hospital de Cruces (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-There Smart Device-2019-001
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Renal Insufficiency, Chronic; Heart Failure; Diabete Mellitus; Diabetes; Nephropathy (Manifestation); Hematuria; Urinary Tract Infections
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure; Diabetes Mellitus; Kidney Diseases; Hematuria; Urinary Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (single arm) (Other): All study participants once enrolled into the study were asked to collect their midstream urine in the designated urine cups. The urine sample was then sent the Lab and tested sequentially; first by the golden standard techniques used by the Lab (first intervention) and by the S-There device (comparative device - second intervention).
  Interventions: Device: Lab Gold Standard; Device: S-There

INTERVENTIONS:
Device: Lab Gold Standard — First intervention (assigned to the "All participants" arm).
Device: S-There — Second intervention (assigned to the "All participants" arm).

SUMMARY:
The objectives of the Clinical Validation Through Analytical Study With Urine Samples to Compare the Effectiveness and Security of an Intelligent Device are:

1.To evaluate the performance of S-There Device in comparison to the golden standard used in the lab.

ELIGIBILITY:
Inclusion Criteria:

* Patients who came to the emergency room, primary care and nephrology unit.

Exclusion Criteria:

* Subject cannot collect urine in receptacle.
* Urinary Catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy to compared device | Through study completion, an average of 1 month
  The primary objective of the study is to evaluate the accuracy of the S-There device compared to the Lab gold standards, for each analyte.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Cruces, Barakaldo, Bizkaia, Spain